CLINICAL TRIAL: NCT01680315
Title: Differences in Physiological Responses of Satiety and Reward After (in)Consistent Calorie Cues.
Brief Title: Calorie Anticipation and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PH2012
Record Dates: First submitted 2012-08-28; First posted 2012-09-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-08

CONDITIONS: Eating Behaviour; Obesity
Keywords: Satiety,; satiation,; anticipation,; food intake
MeSH Terms: conditions — Feeding Behavior; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calorie information (Experimental): Low calorie yogurt
  High calorie yogurt
  with low calorie information sheet
  Interventions: Behavioral: low calorie yogurt; Behavioral: high calorie yogurt
- Calorie information (high) (Experimental): Low calorie yogurt
  High calorie yogurt
  High calorie information sheet
  Interventions: Behavioral: low calorie yogurt; Behavioral: high calorie yogurt

INTERVENTIONS:
Behavioral: low calorie yogurt — all participants consumed twice the low-caloric food (once with the low-calorie information and once with the high-calorie information)
Behavioral: high calorie yogurt — all participants consumed twice the high-caloric food (once with the low-calorie information and once with the high-calorie information)

SUMMARY:
The regulation of our food intake is on the short-term guided by appetite and satiety signals generated by the sight and consumption of food. Food intake is not only regulated by appetite and satiety signals - external cues also play an important role.

It has been observed that food intake and the pleasure derived from consumption is affected by manipulation of the external cues.

The investigators will assess the contribution of food anticipation (calorie information) and actual consumption of a test food (calorie intake) on in satiety responses (such as ghrelin responses, appetite and subsequent food intake). The investigators expect the information on the amount of calories, rather than the actual amount of calories in the food, to predict the ghrelin responses and the subsequent intake of a second meal.

DETAILED DESCRIPTION:
In a randomized cross-over design with 4 conditions, all participants will consume twice the low-caloric food (once with the low-calorie information and once with the high-calorie information) and twice the high-caloric food (again, once with the low-calorie information and once with the high-calorie information) in a randomized order.

ELIGIBILITY:
Inclusion Criteria:

* female
* healthy
* being used to eat breakfast regularly (≥ 5 times a week).

Exclusion Criteria:

* hypersensitivity for the ingredients of the foods under study;
* lack of appetite; following an energy-restricted diet or change in body weight > 5 kg; or
* being a vegan or vegetarian. Participants reported not using products that are artificially sweetened, nor sugar in coffee and/or tea.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Food intake | 60 min (Ad libitum test meal after 1 hr)

SECONDARY OUTCOMES:
Serum concentrations total ghrelin | 60 min (4 samples - every 20 min)

OTHER OUTCOMES:
appetite ratings | 80 min (5 samples - every 20 min)
Serum cortisol concentrations | 60 min (4 samples - every 20 min)

CONTACTS AND LOCATIONS:
Overall Officials: Pleunie Hogenkamp, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

REFERENCES:
- [Derived] Hogenkamp PS, Cedernaes J, Chapman CD, Vogel H, Hjorth OC, Zarei S, Lundberg LS, Brooks SJ, Dickson SL, Benedict C, Schioth HB. Calorie anticipation alters food intake after low-caloric not high-caloric preloads. Obesity (Silver Spring). 2013 Aug;21(8):1548-53. doi: 10.1002/oby.20293. Epub 2013 Apr 13. PMID 23585292